CLINICAL TRIAL: NCT01725633
Title: Phase II Trial of Aerobic Training in Metastatic Breast Cancer
Brief Title: Aerobic Training in Metastatic Breast Cancer
Acronym: Breast Mets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MSKCC 14-170; NCT02239848 (obsolete NCT alias)
Record Dates: First submitted 2011-07-28; First posted 2012-11-14 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Stretching; Nonlinear Aerobic Training; 14-170
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection; Exercise Test

ARMS (2):
- Progressive Stretching Group (Other)
  Interventions: Behavioral: Progressive Stretching Group; Other: Blood draw
- Nonlinear Aerobic Training (Experimental)
  Interventions: Behavioral: Nonlinear Aerobic Training; Other: Blood draw; Other: Cardiopulmonary Exercise Testing (CPET)

INTERVENTIONS:
Behavioral: Progressive Stretching Group — Participants assigned to the progressive stretching group will be provided with a progressive stretching program that matches the aerobic training interventions in terms of program length (16 weeks), social interaction (all sessions will be supervised), and session duration (20-45 minutes/session, ± 10 minutes).
  Arms: Progressive Stretching Group
Behavioral: Nonlinear Aerobic Training — Participants assigned to the nonlinear aerobic training arm will perform no more than 150 minutes per week of structured supervised aerobic training as part of clinical trial participation. Exercise performed outside the structured sessions (i.e., contamination) will be assessed via self-report of exercise behavior using the Godin-Leisure Time Exercise Questionnaire (GLTEQ). For ethical reasons, we will not instruct participants not to exercise outside the structured sessions, but we we will encourage participants to maintain their level of exercise behavior prior to study initiation.
  Arms: Nonlinear Aerobic Training
Other: Blood draw — At Weeks 4, and 8, all participants will have a complete blood count (CBC) test performed.
Other: Cardiopulmonary Exercise Testing (CPET) — At the end of Week 6, participants repeat the CPET in the nonlinear aerobic training group.
  Arms: Nonlinear Aerobic Training

SUMMARY:
This study is being done to examine the safety and feasibility of a supervised progressive exercise program in women diagnosed with metastatic breast cancer. Previous research among women with metastatic breast cancer has shown that some of the treatments commonly used in this population may have an adverse impact on physical fitness levels leading to feelings of fatigue and poor quality of life. Supervised exercise training has been shown to reduce some of these side-effects in women with early-stage breast cancer receiving common cancer treatments. However, it is not known if supervised exercise training is a safe and feasible intervention in women with metastatic breast cancer. This study is designed to find out if supervised exercise training is safe as the patients undergo treatments for metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* MSK histologically confirmed metastatic breast cancer
* Measurable disease (or nonmeasurable bone-only disease) assessed by CT or PET/CT performed as part of standard of care, at the discretion of the attending oncologist in the Breast Medicine Service
* ≥18 years of age;
* Life expectancy >3 months;
* ECOG ≤ 1
* Sedentary, as per the leisure score index (LSI) of the Godin Leisure-Time Exercise Questionnaire (GLTEQ) . Participants who perform regular moderate or vigorous intensity exercise at least 5 days/week, for at least 30 minutes/session, are not eligible
* Able to achieve an acceptable peak baseline CPET, as defined by any of the following criteria:

  1. Achieving a plateau in oxygen consumption, concurrent with an increase in power output;
  2. A respiratory exchange ratio ≥ 1.10;
  3. Attainment of maximal predicted heart rate (HRmax) (i.e., within 10 bpm of age-predicted HRmax [HRmax = 220-Age[years]);
  4. Volitional exhaustion, as measured by a rating of perceived exertion (RPE) ≥ 18 on the BORG scale
* Normal cardiac function (left ventricular ejection fraction ≥50%);
* Medical clearance from attending oncologist indicating no relative contraindications to undergo a symptom-limited cardiopulmonary exercise test and aerobic training intervention;
* Patients with "treated and stable" brain lesions of a duration of ≥ 2 months may be enrolled
* Willing to be randomized to one of the study arms
* Female

Exclusion Criteria:

* Any of the following absolute contraindications to cardiopulmonary exercise testing:

  1. Acute myocardial infarction within 3-5 days of any planned study procedures
  2. Unstable angina
  3. Uncontrolled arrhythmia causing symptoms or hemodynamic compromise;
  4. Recurrent syncope
  5. Active endocarditis;
  6. Acute myocarditis or pericarditis
  7. Symptomatic severe aortic stenosis
  8. Uncontrolled heart failure
  9. Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures
  10. Thrombosis of lower extremities
  11. Suspected dissecting aneurysm
  12. Uncontrolled asthma
  13. Pulmonary edema
  14. Room air desaturation at rest ≤ 85%
  15. Respiratory failure
  16. Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e., infection, renal failure, thyrotoxicosis)
  17. Mental impairment leading to inability to cooperate.
* Any other condition or intercurrent illness that, in the opinion of the investigator, makes the participant a poor candidate for the trial
* Presence of extensive skeletal metastases, defined as more than five (5) sites of bony disease, or any symptomatic site of disease in the spine, hip, or femur. Note that, patients with more than five bony sites may be deemed eligible at the discretion of the attending oncologist.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-12; Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
safety of aerobic training | 2 years
  Safety will be evaluated by the type and prevalence of adverse events during study-related assessments as well as aerobic training and progressive stretching sessions. The NCI Common Terminology Criteria for Adverse Events Version 4.0 (NCI-CTCAE) will be used to grade toxicities during the trial.

SECONDARY OUTCOMES:
feasibility of aerobic training | 2 years
  feasibility will be evaluated by examining several different end points including rates of study eligibility and accrual, etc; however, sample size calculations are based on an integration of aerobic training attendance rate (in the aerobic training group) as well as global trial attrition rates. Together, these end points will be used to determine overall study feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Jones, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Novo RT, Thomas SM, Khouri MG, Alenezi F, Herndon JE 2nd, Michalski M, Collins K, Nilsen T, Edvardsen E, Jones LW, Scott JM. Machine Learning-Driven Phenogrouping and Cardiorespiratory Fitness Response in Metastatic Breast Cancer. JCO Clin Cancer Inform. 2024 Sep;8:e2400031. doi: 10.1200/CCI.24.00031. PMID 39270146
- [Derived] Scott JM, Iyengar NM, Nilsen TS, Michalski M, Thomas SM, Herndon J 2nd, Sasso J, Yu A, Chandarlapaty S, Dang CT, Comen EA, Dickler MN, Peppercorn JM, Jones LW. Feasibility, safety, and efficacy of aerobic training in pretreated patients with metastatic breast cancer: A randomized controlled trial. Cancer. 2018 Jun 15;124(12):2552-2560. doi: 10.1002/cncr.31368. Epub 2018 Apr 6. PMID 29624641
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/